CLINICAL TRIAL: NCT05019339
Title: HomeStyles-2: Shaping HOME Environments and LifeSTYLES to Prevent Childhood Obesity in SNAP-Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB201700192
Record Dates: First submitted 2021-08-11; First posted 2021-08-24 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Healthy Lifestyle; Home Environment Related Disease; Child Behavior; Cognitive Change; Child Obesity; Parenting; Parents; Parent-Child Relations
MeSH Terms: conditions — Child Behavior; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: experimental group and attention control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy HomeStyles (Experimental): Six-week virtual, group nutrition education series using the HomeStyles-2 experimental curriculum administered through SNAP-Ed. This curriculum addresses factors affecting school-aged children's health and nutritional status: inadequate intake of fruits and vegetables, infrequent family meals, excessive consumption of sugar-sweetened beverages, large portion sizes, and irregular breakfast consumption.
  Interventions: Behavioral: Healthy HomeStyles
- Eat Healthy Be Active (Active Comparator): Six-week virtual, group nutrition education series using the Eat Healthy Be Active attention control curriculum administered through SNAP-Ed. This curriculum addresses factors affecting overall health and nutritional status: limiting nutrients of concern (saturated fat, sodium, and added sugars), eating healthy while dining out, eating healthy on a budget, losing weight and keeping it off, understanding nutrition facts labels, and being physically active.
  Interventions: Behavioral: Eat Healthy Be Active

INTERVENTIONS:
Behavioral: Healthy HomeStyles — Comparison of 2 educational interventions
  Arms: Healthy HomeStyles
Behavioral: Eat Healthy Be Active — Comparison of 2 educational interventions
  Arms: Eat Healthy Be Active

SUMMARY:
Childhood obesity prevention efforts are needed in the United States, especially for families with low income. Educating parents and caregivers on simple lifestyle and affordable home environment changes is an effective strategy to improve health outcomes for the entire family. Therefore, the purpose of this study is to determine whether HomeStyles-2, a nutrition education and childhood obesity prevention program for families with children in middle childhood (ages 6 to 11 years), motivates parents to shape their home environments and weight-related lifestyle practices to be more supportive of optimal health and weight status of their children aged 6-11 years more so than those in the control condition. The study will include the experimental group and an attention control group who will engage in a nutrition education program, Eat Healthy Be Active, that is equal in nonspecific treatment effects but does not overlap on topics covered in HomeStyles-2. This study will be implemented in Florida's Supplemental Nutrition Assistance Program-Education (SNAP-Ed) program, which provides nutrition education and obesity prevention supports for individuals with low income who are receiving or eligible for SNAP benefits. Nutrition Educators will be randomized to the experimental or attention control condition, and will lead participants through virtual, group-based nutrition education series. The following data will be collected: sociodemographic characteristics of the participant and child; child and parent health status; parent weight-related cognitions; weight-related behaviors of the participant and child; and weight-related characteristics of the home environment. Enrollment for this study will begin late-2021.

DETAILED DESCRIPTION:
The aim of the HomeStyles-2 for SNAP-Ed families RCT is to determine whether HomeStyles-2 enables and motivates SNAP-Ed parents and child caregivers (e.g., guardians) to shape their home environments and weight-related lifestyle practices to be more supportive of optimal health and weight status of their children aged 6-11 years than those in the control condition. The study will be a two-arm, cluster randomized trial and will follow the CONSORT guidelines extension for cluster trials. Individual counties or groups of small counties operate as a single division with one individual who supervises the SNAP-Ed Nutrition Educators assigned to that division. Every participating division will function as a cluster in the study. Half of the Nutrition Educators in each cluster that choose to participate in the study will be randomized and trained to only deliver the experimental treatment and the other half the control intervention. Eligible participants will be recruited by Nutrition Educators through existing SNAP-Ed community partnerships.

Once identified, eligible individuals will be screened for eligibility, consented, and complete the baseline survey with a trained research assistant over the phone. Participants who complete the baseline survey and meet survey plausibility checks will be enrolled in the study. Their assignment to experimental or attention control condition is dependent upon the Nutrition Educator's random assignment to teach experimental or attention control curriculum. Recruitment materials and the bona fide treatment to be delivered to the attention control group are designed to blind participant assignment to study condition.

Participants will complete a six-week virtual nutrition education program, with each weekly session lasting approximately 30 minutes. Nutrition Educators will conduct the sessions over video conferencing software (e.g., Zoom). Participants will receive intervention materials by mail before the first class of the series and will have electronic access to the materials through a free learning management system. After the six-week virtual nutrition education program, participants will be invited to take the post survey over the telephone with a trained research assistant. Approximately 4 to 10 weeks after participants complete the post survey, they will be invited to take the follow-up survey to assess longer-term intervention effects.

Participant progress through the RCT will be monitored by tracking attendance at each educational session. Trained research assistants and SNAP-Ed staff will be available to answer questions throughout the study. Participants will receive modest stipends that increase in value after they complete each survey.

The HomeStyles-2 experimental group intervention materials (i.e., "Healthy" HomeStyles-2) were designed to be congruent with White House and IOM recommendations for home-centered obesity prevention interventions and critical elements for effective interventions (e.g., interventions are positive, culturally sensitive, supportive of parent-child interaction and child development; develop realistic, effective plans that empower families). HomeStyles-2 for middle childhood intervention materials provide intensive, interactive, fun, non-judgmental opportunities for parents to shape their home environments and lifestyle practices to protect child health. They also promote positive strategies and changes that adults can control in their environments to reduce risk of excessive weight gain in their middle childhood youth. Key factors contributing to childhood obesity that can be suitably addressed in the home environment with middle childhood kids identified for inclusion in the intervention materials were selected using systematic literature reviews and input from experts in childhood obesity prevention. The topics that emerged and will be covered in the SNAP-Ed arm of the study include inadequate intake of fruits and vegetables, infrequent family meals, excessive consumption of sugar-sweetened beverages, large portion sizes, and irregular breakfast consumption. An additional factor was children's limited food preparation skills.

The attention control group will receive a different but bona fide, credible treatment at the same time as the experimental group. The control condition will provide information distinct from the "active" ingredient in the experimental intervention, while still aligning with the description of the study recruitment materials (i.e., to build happier, healthier families) and adhering to the regulations governing educational content of SNAP-Ed programming. The control condition materials are from the SNAP-Ed Eat Healthy, Be Active program and were adapted to match the experimental intervention in number of sessions, length of sessions, 4-page informational guide, goal-setting activity, and incentive items.

To adapt the experimental and control programs for virtual delivery, a Microsoft PowerPoint presentation and script was created for each of the educational sessions. The scripts include suggested questions and opportunities for Nutrition Educators to use to actively engage participants in the session, such as by speaking, typing questions and comments in the chat box, or using emojis to register reactions.

The study survey, "Home Obesogenicity Measure of EnvironmentS"-Families with School-age Kids (HOMES-FSAK), will be used to collect baseline, post, and follow-up data in the HomeStyles-2 RCT. The Social Cognitive Theory along with the key concepts addressed in the HomeStyles-2 guides provided the framework for identification of cognitions, behaviors, and aspects of the home environment to be assessed. The survey will collect sociodemographic characteristics of the participant and child; child and participant health status; parent weight-related cognitions; weight-related behaviors of the parent and child; and weight-related characteristics of the home environment.

ELIGIBILITY:
Inclusion Criteria:

* SNAP-Ed-eligible (i.e., eligible for or receiving SNAP benefits, household income at or below 200% Federal Poverty Guidelines, or living in communities with significant (50% or greater) low-income population)
* Parent or caregiver of a least 1 child aged 6 to 11 years
* Have regular Internet and/or telephone access
* Can read and comprehend English or Spanish
* Reside in study catchment area (i.e., Florida)
* Have not previously participated in nutrition education series using the attention control curriculum

Exclusion Criteria:

* Does not fit inclusion criteria

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Participant weight-related behaviors | Baseline up to follow-up (~4 weeks after post-intervention)
  Participant dietary intake and physical activity behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Karla Shelnutt, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florda, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carman K, O'Neal LJ, Byrd-Bredbenner C, Olfert MD, Shelnutt KP. HomeStyles-2 for SNAP-Ed families with children in middle childhood: Cluster randomized trial protocol. Contemp Clin Trials. 2022 Jun;117:106771. doi: 10.1016/j.cct.2022.106771. Epub 2022 Apr 27. PMID 35489646